CLINICAL TRIAL: NCT01122459
Title: Evaluation of the Effects of Two Types of Fluid in the Recovery From Anaesthesia.
Brief Title: Evaluation of the Effect of Two Types of Fluid in the Recovery From Anaesthesia. Voluven 6% v Hartmanns
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Rotunda Hospital (Other)
Responsible Party: Dr Conan McCaul, Rotunda Hospital/ University College Dublin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RotAnaesFluid1
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2010-05

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Perioperative intravenous fluids
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Hypodermoclysis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hartmanns (Active Comparator): These patients will receive Hartmanns during anaesthesia
  Interventions: Other: fluid administration
- Voluven 6% (Active Comparator)
  Interventions: Other: fluid administration

INTERVENTIONS:
Other: fluid administration — 1.5mls/kg/hr fasting

SUMMARY:
Avoiding nausea and vomiting is one of the most important for patient comfort and satisfaction, and preventing unplanned overnight stays in hospital following surgery. Studies have shown that increased amounts of intravenous fluid during surgery prevent nausea and vomiting after operations. This effect lasted for up to 48 hours after the surgery. Other unpleasant side effects of dehydration that delay recovery including headaches and dizziness can be prevented with fluid treatment during the operation. It is unclear if this effect happens with all types of fluid. The investigators propose to examine the effect of 2 types of intravenous fluids on recovery from anaesthesia. Each group will be given a different fluid while using our usual anaesthetic technique. The investigators will ask questions about nausea and vomiting after surgery (primary outcomes), and other factors relating to patient comfort such as headache and dizziness (secondary outcomes)

DETAILED DESCRIPTION:
Treatment of postoperative nausea and vomiting (PONV) is extremely important for patient comfort and satisfaction after surgery.1 There has been a recent change in emphasis from inpatient to day care surgery and anaesthesia with attendant increased interest in the problem of PONV. The incidence of PONV following day case gynaecologic surgery is 40% to 90%.2,3 Postoperative nausea and vomiting has the potential to cause delays in meeting discharge criteria both from the recovery room to ward, and from the day ward to home. On rare occasions, it may lead to unanticipated overnight hospital admission which leads to an increased emotional cost to the patient and economic cost to the healthcare provider. The efficacy of routine use of prophylactic antiemetics remains controversial.4 Pharmacologic prophylaxis has limited effect and increases the risk of adverse drug effects for the patient in addition to increasing overall cost of care.5,6

Studies suggest that increased crystalloid infusion for day case gynaecologic procedures in healthy patients reduces the incidence of nausea, vomiting and antiemetic use.7,8 The suggested mechanism is an improvement in gastrointestinal mucosal perfusion that mitigates the both the deleterious effects of preoperative fasting and consequent dehydration,9 and those of raised intra-abdominal pressure and surgical manipulation of bowel during laparoscopic procedures. However, excessive fluid administration in major surgery has been shown to have a negative effect on postoperative gastrointestinal function (causing an increased incidence of postoperative ileus) due to bowel oedema.10 It has been demonstrated that colloid causes less bowel oedema than equivalent volumes of crystalloid.11 Moretti et al showed that intraoperative colloid administration reduces PONV and improves the quality of postoperative recovery versus crystalloid solutions.¹² Clearly, there is an optimum perioperative fluid balance to reduce PONV without the risk of additional gastrointestinal side effects.

An arbitrary perioperative fluid load measured in ml.kg-1 does not take account of the individual fasting period and resultant preoperative fluid deficit for each patient, which can vary substantially depending on early or late (morning or afternoon) operating time.

We propose to prospectively examine the effect of intravenous fluids on PONV in a double-blind study, utilizing a standardised anaesthetic technique as normally carried out in this hospital. We hypothesise that replacement of preoperative fluid deficit with colloid will reduce the incidence of PONV versus crystalloid solution. We further propose to examine secondary outcomes relating to patient wellbeing such as headache and dizziness which are symptoms of dehydration.

Healthy patients should not experience any cardiorespiratory effects associated with administration of intravenous fluids to correct dehydration due to preoperative fasting. There may however be subclinical effects which can be detected by sensitive pulmonary function testing. Patients will be asked to perform a simple bedside lung function test before surgery and 2 hours after surgery. This will be done with a portable spirometer (Micromedical Micro Lab Spirometer), which is used routinely in our anaesthesia preoperative assessment clinic to evaluate lung function. Forced expiratory volume in the first second (litre) (FEV1), forced vital capacity (litre) (FVC) and peak flow rates (l/min) will be measured at a 45 degree position of recumbency. The best of three attempts will be chosen for further analysis as recommended by the British Thoracic Society.

Methods

LOCATION · Rotunda Hospital, operating theatres, recovery room and gynaecology ward

STUDY DESIGN

· Prospective, randomised, double-blind

INCLUSION CRITERIA

* ASA I-II female patients
* Age 18-45 years
* Undergoing minor elective gynaecological surgery (elective laparoscopy)

EXCLUSION CRITERIA

* Age <18 or > 45
* Cardio-respiratory disease
* Excessive intraoperative blood loss
* Obesity: BMI >30
* Relevant drug allergy to medication used in the protocol

INFORMED WRITTEN CONSENT · Informed written consent will be obtained from all patients (see appendix 1)

RANDOMISATION

· Patient group will be determined by randomisation with a computer program random number generator

GROUPS

* Patients will be allocated to one of two groups according to randomisation
* Group 1 will receive 1.5 ml.kg.hr-1 of fasting time of intravenous Hartmann's solution perioperatively (Crystalloid solution)
* Group 2 will receive 1.5 ml.kg.hr-1 of fasting time of intravenous Voluven® (6% Hydroxy Ethyl Starch) solution perioperatively (Colloid solution)

BLINDING

* All fluid administration will be completed in theatre
* Neither the patient or the investigator will be aware of group assignment

ANAESTHETIC TECHNIQUE The anaesthetic technique will be standardised as follows: Intravenous access will be obtained after local anaesthetic infiltration of the skin. Once the fluid has been started all patients will undergo a standardised induction of anaesthesia, consisting of Fentanyl 1.5 mcg.kg-1, Propofol 2-3 mg.kg-1 and Atracurium 0.35 mg.kg-1 to facilitate airway control. All patients will be mechanically ventilated via a laryngeal mask airway LMA Supreme™ to maintain isocapnia with tidal volume (Vt) 4-6 ml.kg-1, maximum airway pressure (P max) 30 cm H2O and a positive end expiratory pressure (PEEP) of 5 cm H2O. Anaesthesia will be maintained with Sevoflurane 1-3% in a mixture of O2 and air to achieve a FiO2 of 0.5. Muscle relaxation will be antagonised with Neostigmine 2.5 mg and Glycopyrrolate 0.5 mg at the end of surgery. Before discontinuation of anaesthesia, each patient will receive rectal Diclofenac 100mg and 1000mg Paracetamol i.v.

Postoperative care will also be standardised. Patients complaining of pain will be given 25 mcg of Fentanyl intravenously as required (in PACU), Pethidine 50mg intramuscularly or simple oral analgesics (Paracetamol/Codeine 500-1000mg/8-16mg) every 6 hours in the ward area. Rescue antiemetics in the form of boluses of Ondansetron 4mg intravenously (to a maximum total dose of 16mg) and Cyclizine 50mg intramuscularly every 8 hours can be given. Patients will be prescribed oral Paracetamol/Codeine 500-1000mg/8-16mg every 6 hours and Diclofenac 50mg every 8 hours to take at home if required.

MEASUREMENTS (assessed by a single data collector @ 30 mins, 2 hours, 24 hours and 48 hours postoperatively)

1. Nausea: using a standard verbal analogue scale (VAS 0 - 10)
2. Vomiting: Y/N, number of episodes
3. Rescue antiemetics administered
4. Dizziness: Y/N
5. Sore throat: Y/N
6. Headache: Y/N
7. Wellbeing: assessment of general wellbeing on a scale from 0 - 10
8. Pulmonary Function Tests

TREATMENT OF DATA The data will be collected by a single investigator at the specified time points and documented on a patient data collection sheet (see appendix 2). Once data collection is complete, all data of the patient sheets will be transferred onto a spreadsheet and anonymised.

USE OF DATA The data will be presented at a national or international meeting and in peer-reviewed medical journals.

STORAGE OF DATA All data will be stored for five years and only Dr. Conan McCaul and Dr. Ivan Hayes will have access to them.

STATISTICAL PROCEDURES Statistics will be performed using a standard statistical program (Sigma Stat, Jandel Scientific). Demographic data will be analysed using Student's t-test or Fisher's exact test as appropriate. Repeated measures ( VAS scores) will be analysed by repeated measures analysis of variance with further paired comparisons at each time interval performed using the t-test, with corrections for multiple comparisons where appropriate. Categorical data will be analysed using χ² analysis or the Fisher's exact test where applicable. Normally distributed data will be presented as means +/-SEM, non-normally distributed data will be presented as medians +/- quartiles (interquartile range), and categorical data will be presented as raw data and as frequencies.

SAMPLE SIZE Postoperative nausea and vomiting incidence from day case laparoscopic gynaecologic procedures (primary outcome) both with and without single agent antiemetic prophylaxis varies from 40 -90%.2,3,7 To detect a clinically significant difference of 25% reduction in mean nausea scores based on a PONV incidence of 40% without antiemetic prophylaxis, we calculate a sample size of 60 patients per group (a = 0.05, β = 0.2).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiology classification 1 & 2
* Minor laparoscopic gynaecological surgery
* Age 18-45

Exclusion Criteria:

* Age <18 or > 45
* Cardio-respiratory disease
* Obesity: BMI >30
* Relevant drug allergy to medication used in the protocol

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Incidence of nausea and vomiting | 120 mins

SECONDARY OUTCOMES:
Incidence of Headache | 30 mins
Incidence of headache | 120 mins
Incidence of headache | 24 hours
Incidence of headache | 48 hours
Incidence of nausea and vomiting | 30 mins
Incidence of nausea and vomiting | 24 hours
Incidence of nausea and vomiting | 48 hours
Incidence of sore throat | 30 mins
Incidence of sore throat | 120mins
Incidence of sore throat | 24 hours
Incidence of sore throat | 48 hours
Incidence of dizzyness | 30 mins
Incidence of dizzyness | 120 mins
Incidence of dizzyness | 24 hours
Incidence of dizzyness | 48 hours
Verbal analogue scale of general wellbeing | 30 mins
Verbal analogue scale of general wellbeing | 120 mins
Verbal analogue scale of general wellbeing | 24 hours
Verbal analogue scale of general wellbeing | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Rotunda Hospital, Dublin, Dublin, Ireland